CLINICAL TRIAL: NCT06024018
Title: Efficacy of High Intensity Electromagnetic Body Shaping in Obese Men
Brief Title: Effect of High Intensity Electromagnetic Body Shaping on Profile of Metabolism in Obese Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003755
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Central Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first group (Experimental): thirty obese males (30 males) will undergo dietary caloric restriction and will be instructed to walk 10,000 continuous steps every day using the pedometer application for 3 months. Also they will undergo high intensity electromagnetic technique (40 minutes for every session) on abdomen of males which will be 3 sessions per week for 3 months
  Interventions: Device: high intensity electromagnetic technology device, diet restriction, and walking
- second group (Active Comparator): thirty obese males (30 males) will undergo dietary caloric restriction and will be instructed to walk 10,000 continuous steps every day using the pedometer application for 3 months.
  Interventions: Behavioral: diet restriction and walking

INTERVENTIONS:
Device: high intensity electromagnetic technology device, diet restriction, and walking — thirty obese males (30 males) will undergo dietary caloric restriction and will be instructed to walk 10,000 continuous steps every day using the pedometer application for 3 months. Also they will undergo high intensity electromagnetic technique (40 minutes for every session) on abdomen of males which will be 3 sessions per week for 3 months
  Arms: first group
Behavioral: diet restriction and walking — thirty obese males (30 males) will undergo dietary caloric restriction and will be instructed to walk 10,000 continuous steps every day using the pedometer application for 3 months.
  Arms: second group

SUMMARY:
high intensity focused electromagnetic technology's secondary effects are observed in the fat (adipose). within 8 h of a treatment session, apoptotic levels in adipose increased 91.7%.8 In addition, after the application of the high intensity electromagnetic technique, there is an increase in the rapid release of free fatty acids, so it can be used in weight loss

DETAILED DESCRIPTION:
sixty obese males will be grouped to: first group (30 males) and second group (30 males). first and second groups will undergo dietary caloric restriction (i.e low calorie diet) and will be instructed to walk 10,000 continuous steps every day using the pedometer application for 3 months. only the first group will will undergo high intensity electromagnetic technique on abdomen of males which will be 3 sessions per week for 3 months

ELIGIBILITY:
Inclusion Criteria:

* men with central obesity
* BMI 30-34.9 kg/m2

Exclusion Criteria:

* metabolic /cardiovascular, pulmonary illnesses, musculoskeletal/neurological illness, autoimmune/psychological illnesses

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
subcutaenous abdominal fat thickness | 12 weeks
  it will be measured using ultrasonography

SECONDARY OUTCOMES:
visceral abdominal fat thickness | 12 weeks
  it will be measured using ultrasonography
body mass index | 12 weeks
  it will be measured at morning with empty stomach and bladder
waist circumference | 12 weeks
  it will be measured using inelastic tape
cortisol | 12 weeks
  it is a stress hormone
high density lipoprotein | 12 weeks
  it will be measured in serum
low density lipoprotein | 12 weeks
  it will be measured in serum
triglycerides | 12 weeks
  it will be measured in serum
cholesterol | 12 weeks
  it will be measured in serum
appearance of abdomen subscale of Body Q questionnaire | 12 weeks
  BODY-Q provides a set of scales focusing on topics that are relevant to weight
health related-quality-of-life subscale of Body Q questionnaire | 12 weeks
  it provids questions related to body image , physical function , psychological function , sexual function
eating related concerns subscale of Body Q questionnaire | 12 weeks
  it provids questions related to eating behavior , expectations weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Study Director — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt